CLINICAL TRIAL: NCT01545349
Title: Double Blind Randomized Controlled Trial to Evaluate the Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) Versus Placebo in Elderly Subjects Receiving Live Attenuated Influenza Vaccine
Brief Title: Safety of Lactobacillus Rhamnosus GG Versus Placebo in Elderly Subjects Receiving Live Attenuated Influenza Vaccine
Acronym: LAIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patricia L. Hibberd (Other)
Responsible Party: Sponsor-Investigator, Patricia L. Hibberd, Chief, Division of Global Health; Department of Pediatrics, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2011 P 002849
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Healthy; Influenza
Keywords: LGG; Immune response; Influenza vaccine; Elderly; Healthy; Microbiome
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG (Experimental): Lactobacillus rhamnosus GG (LGG) containing 1x10^10 LGG per capsule will be given to subjects with verbal and written instructions at the baseline visit. Capsules are to be taken orally twice a day on an outpatient basis.
  Interventions: Biological: Lactobacillus rhamnosus GG ATCC 53103 (LGG); Biological: Live attenuated influenza vaccine
- Placebo (Placebo Comparator): Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day on an outpatient basis.
  Interventions: Biological: Placebo; Biological: Live attenuated influenza vaccine

INTERVENTIONS:
Biological: Lactobacillus rhamnosus GG ATCC 53103 (LGG) — Study drug capsules (1x10^10 LGG/capsule) are to be taken orally twice a day every day on an outpatient basis for 28 days
  Other Names: Culturelle
  Arms: LGG
Biological: Placebo — Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day on an outpatient basis for 28 days.
  Arms: Placebo
Biological: Live attenuated influenza vaccine — 0.2 mL pre-filled, single use intranasal spray
  Other Names: FluMist

SUMMARY:
This is a Phase I, randomized controlled trial to evaluate the safety of Lactobacillus rhamnosus GG (LGG) versus placebo in elderly subjects receiving the live attenuated influenza vaccine. Lactobacilli are part of the normal flora of the intestine. LGG is one of several strains of Lactobacilli that is used as a probiotic or microorganism administered to confer "health benefits". Our research is focused on studying the possible therapeutic effects of LGG. The study hypotheses are:

1. LGG or placebo administered twice daily will be safe and well tolerated in elderly subjects who have just received the live attenuated influenza vaccine,
2. The immune response to the influenza vaccine at day 21, 28, and 56 will be higher in the LGG group than the placebo group,
3. The diversity of the microbiota in nasopharyngeal and stool specimens at day 21, 28, and 56 will be greater in the LGG group than the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-80 years
2. Willing to complete the informed consent process
3. Able and willing to participate for the planned duration of the study, including availability for follow-up telephone contact
4. Is community dwelling for the past two years
5. Has received routine physical in the past two years
6. Has no new chronic conditions in the past two years
7. Identifies a primary care clinician
8. Has received recommended preventive services (Task Force for Clinical Preventive Services) for vaccination and cancer prevention/detection, e.g.:

   * Pneumococcal vaccination
   * Mammography
   * Screening colonoscopy for colon cancer
9. Willing to comply with protocol and report on compliance and side effects during the study period
10. Informed consent obtained and signed prior to screening

Exclusion Criteria:

1. Vaccination with any vaccine within the one month period prior to study enrollment or intent to receive any other vaccine during the study period, other than TIV in fall 2012
2. History of hypersensitivity to any influenza vaccine components including eggs, egg proteins, gentamicin, gelatin or arginine
3. History of avoidance of egg and/or egg-based products for any reason, unless they have previously received TIV or LAIV without hypersensitivity
4. History of Guillain-Barre syndrome
5. Acute febrile illness within the week prior to LAIV immunization - immunization deferred until illness resolved
6. Consumption of supplements or food products containing LGG or probiotics for 28 days prior to the start of the study or consumption of yogurt that has the "live and active" cultures seal
7. Known or suspected allergies to probiotics, Lactobacillus, microcrystalline cellulose, gelatin or antibiotics that may be used to treat LGG bacteremia or infection (i.e., subject able to tolerate at least 2 of the following regimens - Ampicillin or other beta lactam antibiotic, and Clindamycin, and Moxifloxacin)
8. Received oral or parenteral antibiotics within 4 weeks of enrollment or prescribed antibiotics on the day or enrollment
9. Drug or alcohol abuse, defined as the continued use of alcohol despite the development of social, legal, or health problems, within the previous 12 months
10. Hospitalization, major surgery or endoscopy within the last 3 months
11. Scheduled hospital admission or surgery within 3 months of enrollment
12. Resident of a nursing home or rehabilitation center
13. Close and/or household contact with severely immunocompromised persons (e.g., transplant recipients, cancer patients)
14. Receipt of any of the following medications within the specified time frame:

    * Antiviral agents for influenza A and B in the prior 2 weeks (anti-influenza medications are unlikely to be needed after LAIV immunization since LAIV will be administered at the end of the influenza season, but should be prescribed if clinically indicated)
    * Immune Globulin within the prior 6 months
    * Immune modulating drugs such as Belimumab, azathioprine, mercaptopurine, methotrexate, hydroxychloroquine or leflunomide at any time or any oral or parenteral corticosteroid in the prior 12 months
    * Fingolimod at any time
    * Salicylates at doses higher than 163 mg/day for primary prevention of myocardial infarction. (Reye's Syndrome in adults is extremely rare - to our knowledge the oldest reported patient was aged 61 and as of 1989 when Reye Syndrome was more common, it had only been reported in 25 adults. In addition, increasing numbers of adults are being placed on low dose aspirin for primary and secondary prevention of cardiovascular disease, some of whom may also have influenza, but there has been no increase in reports or Reye's Syndrome in adults.)
15. Presence of any of the following:

    * Grade 2 or higher abnormal vital signs or abnormalities on physical exam during screening or presence of any wheezing on physical exam at baseline
    * Indwelling catheter or implanted hardware/prosthetic device or feeding tube
    * Current or within the last 2 years, any episode of bowel leak, acute abdomen, diverticulitis, colitis, bloody bowel movements or peptic ulcer disease, including any surgical procedure or current prescription medications for any of these conditions
    * Current or within the last four weeks, active bowel disease such as an episode of infectious or non-infectious diarrhea, constipation or vomiting lasting more than 12 hours or current prescription medications for any of these conditions
    * Any history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, history of gastrointestinal tract cancer or metastasis or inflammatory bowel disease or current prescription medication for any of these conditions
    * Any history of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease
    * Underlying structural heart disease such as abnormal native heart valve or congenital abnormality, previous history of endocarditis or valve replacement, Stage IV congestive heart failure or chronic cardiovascular conditions (except hypertension)
    * History of peripheral vascular disease or stroke
    * Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy, neutrophil count < 500/mm3, or an anticipated drop in the neutrophil count to < 500/mm3 during the 56 days post LAIV vaccination or active or planned chemotherapy or radiotherapy
    * History of collagen vascular or autoimmune disease
    * History of renal disease
    * History of chronic obstructive pulmonary disease or asthma
    * History of neurologic or neuromuscular diseases
    * History of hematologic diseases
    * Diabetes or thyroid disease or metabolic disorder
    * Active tuberculosis (TB), defined as undergoing a work up for suspected active TB infection or currently on treatment for active TB or scheduled for tuberculin test in the next 4 weeks
    * Fever or acute illness or nasal congestion during the baseline visit (LAIV administration)
16. Positive drug or alcohol testing at screening or positive breathalyzer at baseline or an unwillingness to undergo drug and alcohol testing
17. Abnormal laboratory tests defined as any of the following:

    * White blood cell (WBC)< 3.3 or > 12.0 K/microliters
    * Neutrophil < 500/mm3
    * Platelets < 125 K/microliter
    * Hemoglobin males: < 12.0 g/dL; females: < 11.0 g/dL
    * Creatinine > 1.8 mg/dL
    * Blood urea nitrogen (BUN) > 27 mg/dL
    * Aspartate aminotransferase (AST) > 1.25 ULN
    * Alanine aminotransferase (ALT) > 1.25 ULN
    * Alkaline phosphatase > 1.25 ULN
    * Bilirubin (total) > 1.5 ULN
    * Glucose (non-fasting) > 126 mg/dL
    * Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody
18. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the subject participating in the study or would make it unlikely the subject could complete the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events that are possibly or probably related to administration of LGG | Subjects will be followed from the study start through the end of the 2012-2013 influenza season (as defined by CDC) with an anticipated average for most subjects of 13 months
  Adverse events will be detected during study visits with standardized questionnaires, medical history, vital signs, physical examinations, laboratory tests and review of subject diaries as well as between study visits on telephone calls based on responses to adverse event questionnaires. Additionally, subjects are encouraged to call the PI or study staff at any time if they are experiencing an adverse event.

SECONDARY OUTCOMES:
Anti-influenza systemic immune response (HAI, MN titers and IgA titers) | Baseline through day 56 post LAIV vaccination
  HAI, MN titers and IgA titers will be measured at baseline and on days 21, 28, 56 post LAIV vaccination
Anti influenza mucosal immune response (IgA titers) | Baseline through day 56 post LAIV vaccination
  IgA levels will be measured at baseline, and days 21, 28 and 56 post LAIV immunization
Richness and microbial diversity in nasopharyngeal and stool specimens | Baseline through day 56 post LAIV vaccination
  Measure of the richness and microbial diversity in nasopharyngeal and stool specimens using pyrosequencing
Anti influenza systemic immune response post TIV vaccination | Fall 2012 - prior to and 28 days post TIV vaccination
  Anti influenza systemic immune response (HAI and MN titers) will be measured before and 28 days after TIV immunization in the fall 2012.
Occurence of influenza-like illness during 2012-2013 influenza season | Baseline through the end of the 2012-2013 influenza season (anticipated average of 13 months)
  Subjects will telephoned every month after receiving the TIV vaccination in the fall of 2012, through the end of the 2012-2013 influenza season, to determine if they have an influenza-like illness. They will also be asked to keep a study diary if they experience any influenza-like symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States